CLINICAL TRIAL: NCT02931409
Title: Intraoperative PEEP Optimization: Effects on Postoperative Pulmonary Complications and Inflammatory Response. A Double-center, Prospective, Randomized Controlled Trial
Brief Title: Intraoperative PEEP Optimization: Effects on Postoperative Pulmonary Complications and Inflammatory Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Péterfy Sándor Hospital (Other)
Collaborators: Szeged University (Other)
Responsible Party: Principal Investigator, Dr. Zoltán Ruszkai, Deputy Head of Department of Anaesthesiology and Intensive Care, Péterfy Sándor Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21586-4/2016/EKU; CO-338-045 (Other: Péterfy Sándor Hospital Scientific Research Ethics Committe); 149/2016-SZTE (Other: University of Szeged Human Investigation Review Board)
Record Dates: First submitted 2016-10-05; First posted 2016-10-13 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Complications; Inflammatory Response
Keywords: Positive end-expiratory pressure; Static pulmonary compliance; Lung Protective Ventilation; Radical cystectomy and urinary diversion; Postoperative pulmonary complications; Procalcitonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal PEEP (Experimental): Patients submitted to general anesthesia and open radical cystectomy and urinary diversion (20 subjects) will be submitted an alveolar recruitment maneuver using the sustained airway pressure by the CPAP method, applying 30 cmH2O PEEP for 30 seconds followed by a decremental PEEP titration procedure directed by static pulmonary compliance (Cstat). During PEEP titration procedure PEEP will be decreased from 14 cmH2O by 2 cmH2O every 4 minutes, until a final PEEP of 6 cmH2O. Optimal PEEP is considered as a PEEP value resulting the highest possible Cstat measured by ventilator. After PEEP titration procedure a lung protective mechanical ventilation will be performed using optimal PEEP and low tidal volumes (6 mL/Kg IBW).
  Interventions: Procedure: Optimal PEEP
- Standard PEEP (Active Comparator): Patients submitted to general anesthesia and open radical cystectomy and urinary diversion (20 subjects) will be submitted an alveolar recruitment maneuver using the sustained airway pressure by the CPAP method, applying 30 cmH2O PEEP for 30 seconds followed by a standard lung protective mechanical ventilation using a PEEP value of 6 cmH2O and low tidal volumes (6 mL/Kg).
  Interventions: Procedure: Standard PEEP

INTERVENTIONS:
Procedure: Optimal PEEP — Optimal PEEP determined by Cstat during PEEP titration procedure.
  Arms: Optimal PEEP
Procedure: Standard PEEP — Lung protective mechanical ventilation applying a PEEP value of 6 cmH2O
  Arms: Standard PEEP

SUMMARY:
The purpose of this prospective randomized controlled trial is to determine the effects of intraoperative lung protective mechanical ventilation using an individual optimal PEEP value on postoperative pulmonary complications and inflammatory response. A total number of 40 patients undergoing open radical cystectomy and urinary diversion will be enrolled and randomized into two groups. Standard lung protective ventilation using a PEEP of 6 cmH2O will be performed in control group and an optimal PEEP value determined during a static pulmonary compliance (Cstat) directed PEEP titration procedure will be applyed in study group. Low tidal volumes (6mL/Kg IBW) and a fraction of inspired oxygen (FiO2) of 0.5 will be applyed in both groups. Procalcitonin kinetics will be monitored during and after surgery until the third postoperative day as well as postoperative pulmonary complications. Clinical condition and extrapulmonary complications will be evaluated by the Sequential Organ Failure Assessment (SOFA) Score and in-hospital stay, 28-days and in-hospital mortality will also be followed.

DETAILED DESCRIPTION:
Patients undergoing general anesthesia and mechanical ventilation during major abdominal surgery commonly develop pulmonary atelectasis or even hyperdistension of the lungs can occur leading to adverse consequences either intraoperatively or postoperatively. Lung protective ventilation (LPV, PEEP = 6 cmH2O, TV = 6 mL/Kg IBW and regular recruitments) during the intraoperative period can reduce the risk of ventilator induced lung injury (VILI) and prevent the formation of pulmonary atelectasis.

In our investigator-initiated, double-center, single-blinded, prospective, randomized, controlled clinical trial a total number of 40 patients with bladder cancer undergoing open radical cystectomy and urinary diversion (ileal conduit or orthotopic bladder substitute) will be enrolled and randomized into two groups. Standard lung protective mechanical ventilation with the use of 6 cmH2O of PEEP and low tidal volumes (6mL/Kg IBW), a fraction of inspired oxygen (FiO2) of 0.5 and a respiratory rate to maintain an end tidal carbon dioxide (ETCO2) between 35-40 mmHg will be performed in control group, and a strategy of lung protective mechanical ventilation applying an optimal, individual PEEP determined by static pulmonary compliance (Cstat) directed PEEP titration procedure will be performed in study group.

During preoperative assessment, respiratory failure risk index (RFRI) will be recorded and informed consent will be obtained. Regarding to the protocol, a central vein catheter will be placed on the day before surgery, serum procalcitonin (PCT) level will be measured and a chest X-ray examination will be performed.

Before induction of anesthesia, an epidural catheter and an arterial canula for invasive blood pressure monitoring will be inserted. Immediately after induction of anesthesia and orotracheal intubation, all patients will be submitted to an alveolar recruitment maneuver (ARM) using the sustained airway pressure by the CPAP method, applying 30 cmH2O PEEP for 30 seconds. After ARM PEEP will be set to 6 cmH2O in the control group ("standard PEEP") and LPV will be performed. In the study group ("optimal PEEP") PEEP will be set to 14 cmH2O and a Cstat directed decremental PEEP titration procedure will be performed (every 4 minutes PEEP will be decreased by 2 cmH2O, until a final PEEP of 6 cmH2O) to determine the best individual PEEP. During surgery ARM will be repeated and arterial and central vein blood gas samples (ABGs, CVBGs) will be evaluated every 60 minutes. PCT levels will be measured 2, 6, 12, 24, 48 and 72 hours after surgical incision.

After extubation, patients will be addmitted to the Department of Anesthesiology and Intensive Care. ABGs and CVBGs will be collected and evaluated, PaO2/FiO2 and dCO2 will be calculated every 6 hours until 72 hours after surgery. On the first postoperative day chest X-ray will be performed and repeated on the following days if developing of pulmonary complications were suspected. Continuous epidural analgesia will be introduced, and evaluated effective if numeric pain rating scale point would be lower than 3 points.

During postoperative care continuous intraabdominal pressure (IAP) monitoring via a direct intraperitoneal catheter placed before closure of the abdominal wall will be performed to eliminate bias caused by the elevation of intraabdominal pressure.

Patients' clinical progress and secondary endpoints will be monitored by daily SOFA Scores, laboratory and physical examinations.

During follow-up period in-hospital stay, 28-days and in-hospital mortality will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bladder cancer undergoing radical cystectomy and urinary diversion (ileal conduit or orthotopic bladder substitute)

Exclusion Criteria:

* Age < 18 years
* ASA grade IV
* History of severe chronic obstructive pulmonary disease (COPD, GOLD grade III or IV)
* History of severe or uncontrolled bronchial asthma
* History of severe restrictive pulmonary disease
* Pulmonary metastases
* History of any thoracic surgery
* Need for thoracic drainage before surgery
* Renal replacement therapy prior to surgery
* Congestive heart failure (NYHA grade III or IV)
* Extreme obesity (BMI > 35 Kg/m2)
* Lack of patient's consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Pulmonary Complications | 72 hours
  New infiltrates or atelectasis on chest X-ray, abnormal breathing sounds on auscultation, excessive bronchial secretions, unexplained fever, respiratory failure defined as PaO2/FiO2 < 300 or need for non-invasive or invasive ventilatory support.
Procalcitonin Kinetics | 72 hours
  Serum procalcitonin levels during and after surgery.

SECONDARY OUTCOMES:
Incidence of Circulatory Failure | 28 days
  Severe hypotension, arrhytmias, decreased cardiac output, severe metabolic acidosis, congestive heart failure, acute coronary syndrome, pulmonary embolism and cardiac arrest.
Incidence of Gastrointestinal Dysfunctions | 28 days
  Constipation or ileus, anastomotic leakage and need for urgent reoperation, disorders of liver function.
Incidence of Renal Dysfunction | 28 days
  RIFLE Criteria
Incidence of Hematologic and Coagulation Disorders | 72 hours
  Severe bleeding and/or coagulopathy
Infection | 28 days
  Any infections except from pneumonia.

OTHER OUTCOMES:
ICU days | 28 days
  Defined as a period from the first postoperative day until emission from the ICU.
In-hospital Stay | 28 days
  From the day of surgery until emission from hospital.
Mortality | 28 days
  In-hospital and 28 days mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Molnár, Prof, MD, PhD, DEAA, Study Director — University of Szeged, Faculty of Medicine, Department of Anaesthesiology and Intensive Therapy; Zoltán Ruszkai, MD, Principal Investigator — Péterfy Sándor Hospital, Department of Anaesthesiology and Intensive Care
Locations (2):
- Hungary (2):
  - University of Szeged, Faculty of Medicine, Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye
  - Péterfy Sándor Hospital, Budapest, Pest County

IPD SHARING:
Plan to Share IPD: No
IPD are not relevant in terms of results.

REFERENCES:
- [Derived] Ruszkai Z, Kiss E, Laszlo I, Bokretas GP, Vizseralek D, Vamossy I, Surany E, Buzogany I, Bajory Z, Molnar Z. Effects of intraoperative positive end-expiratory pressure optimization on respiratory mechanics and the inflammatory response: a randomized controlled trial. J Clin Monit Comput. 2021 May;35(3):469-482. doi: 10.1007/s10877-020-00519-6. Epub 2020 May 9. PMID 32388650
- [Derived] Ruszkai Z, Kiss E, Laszlo I, Gyura F, Surany E, Bartha PT, Bokretas GP, Racz E, Buzogany I, Bajory Z, Hajdu E, Molnar Z. Effects of intraoperative PEEP optimization on postoperative pulmonary complications and the inflammatory response: study protocol for a randomized controlled trial. Trials. 2017 Aug 11;18(1):375. doi: 10.1186/s13063-017-2116-z. PMID 28800778